CLINICAL TRIAL: NCT04794946
Title: Safety and Efficacy of a Non-replicating ChAdOx1 Vector Vaccine AZD1222 (COVISHIELD), for Prevention of COVID-19 in Patients With Liver Cirrhosis - A Pilot Study
Brief Title: Safety and Efficacy of a Non-replicating ChAdOx1 Vector Vaccine AZD1222 (COVISHIELD), for Prevention of COVID-19 in Patients With Liver Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-COVID-05
Record Dates: First submitted 2021-03-08; First posted 2021-03-12 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-03

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liver Cirrhosis (Experimental): Evidence of liver cirrhosis established during the clinical investigations and/or hospital stay, as evidenced by clinical, endoscopic, radiological and/or histological criteria.
  Interventions: Biological: Covishield
- Non Liver Cirrhosis (Healthy Control) (Active Comparator): No major respiratory, cardiac comorbid illnesses or malignancy or immunosuppressed state
  Interventions: Biological: Covishield

INTERVENTIONS:
Biological: Covishield — 2 IM doses (0.5 mL) of AZD1222(Covishield) at Day 0 and after 6-8 weeks of first dose (Day 42-56 days). This schedule will be followed for the first 100 participants, following which vaccination schedule as per the prevailing Government protocols shall be followed as a part of Adaptive Clinical Trial.

SUMMARY:
COVID-19 pandemic, caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), had caused widespread impact on health, including substantial mortality among those with pre-existing health conditions including cirrhosis. Patients with liver cirrhosis are at increased risk of severe disease and death from the virus infection that causes COVID-19 and are therefore a priority for immunization, should an efficacious vaccine be developed. Currently, there are no specific treatments available against COVID-19 and cirrhosis patients are a priority group for vaccination.

DETAILED DESCRIPTION:
* Study population: Group 1: Liver Cirrhosis Group 2: Control Group (Healthy controls)
* Study design: A Single Centre, Pilot Study,Adaptive Clinical Trial
* Study period: 1 year, Enrolment Period: Mar 2021 to Aug 2021
* Sample size with justification:

Study is being conducted as a pilot study. First 100 participants will be enrolled in both the groups. However a preliminary analysis will be done after enrollment of 50 participants in each group. Study is being conducted as a Adaptive Clinical Trial.

* Intervention:

  2 IM doses (0.5 mL) of AZD1222(Covishield) at Day 0 and after 6-8 weeks of first dose (Day 42-56 days). This schedule will be followed for the first 100 participants, following which vaccination schedule as per the prevailing Government protocols shall be followed as a part of Adaptive Clinical Trial.
* Monitoring and assessment:

SARS CoV2 serum IgG Levels and neutralizing antibody titers:

The blood samples at baseline (pre first dose), day 28 (4 weeks/28 days after first dose and just before second dose), 8 weeks (or 4 weeks after second dose), 16 weeks (or 12 weeks after second dose), 28 weeks (or 24 weeks after second dose), 40 weeks (or 36 weeks after second dose) and 52 weeks ( or 48 weeks after second dose) Post vaccination will be screened for anti-SARS-CoV-2 IgG by commercially available chemiluminescent immunoassays (CLIA) SARS-CoV-2 IgG (Ortho Clinical Diagnostics, Raritan, NJ, USA)on VITROS ECi/ECiQ/3600 automated instrument. Results will be expressed as reactive with Serum/cut off ratio ≥ 1, and non-reactive with < 1 S/Co ratio.

All reactive samples will be further processed to measure the neutralizing antibody titer utilizing a surrogate virus neutralization test ELISA based commercial assay (sVNT)(GenScript cPass™ SARS-CoV-2 Neutralization Antibody Detection Kit) to look for neutralizing antibody response to the spike protein of the virus.

Real Time PCR for SARS CoV-2 infection:

A diagnosis of SARSCoV-2 infection will be confirmed by performance of Real Time reverse transcriptase polymerase chain reaction (RT-PCR) on the combined nasopharyngeal and oral swab collected in Viral transport medium and by detection of at least 2 specific gene targets of the SARS CoV-2 virus (E and RdRP genes).

Primary IFN-γ ELISPOT assay. The blood samples at baseline (pre first dose), day 28 (4 weeks/28 days after first dose and just before second dose), 8 weeks (or 4 weeks after second dose), 16 weeks (or 12 weeks after second dose), 28 weeks (or 24 weeks after second dose), 40 weeks (or 36 weeks after second dose) and 52 weeks ( or 48 weeks after second dose) will be collected. Primarily, cellular responses will be assessed using an ex-vivo interferon-γ enzyme-linked immunospot (ELISpot) assay to enumerate antigen-specific T cells. In brief, PBMCs will be isolated from whole blood by density gradient centrifugation, immediately cryopreserved in 90% fetal bovine serum and 10% dimethyl sulfoxide, and transferred to liquid nitrogen for storage.

IFN-γ ELISPOT assays will be performed using cryopreserved PBMC. Briefly, unfractionated PBMC will be thawed, resuspended at a concentration of 1 × 106 cells/ml in DMEM medium, and will be plated at 100 μl/well (1 × 105 cells/well) in 96-well, nitrocellulose-backed plates (Millipore Corp, Bedford, MA) previously coated with a PBS solution of anti-IFN-γ monoclonal antibody (1-D1K, 5 μg/ml; Mabtech Technologies, Nacka, Sweden). Along with negative control as, different cell stimuli (PMA; phytohemagglutinin 1 μg/ml and Ionomycin ) will be used in as positive controls., Plates will then incubated at 37°C for 40 h, and then will be harvested and read in ELISPOT reader. A vaccine-induced response will be defined as a ≥3-fold increase over the baseline response to the individual epitope peptide.

T cells Functionality:

The blood samples at baseline (pre first dose), day 28 (4 weeks/28 days after first dose and just before second dose), 8 weeks (or 4 weeks after second dose), 16 weeks (or 12 weeks after second dose), 28 weeks (or 24 weeks after second dose), 40 weeks (or 36 weeks after second dose) and 52 weeks ( or 48 weeks after second dose) Immune response measurements will be assessed using peripheral blood mononuclear cells (PBMC) obtained at all time points.

To investigate the CD4 and CD8 T cell functionality PBMCs will be cultured in 96 well plate in RPMI media containing 10% FBS, with or without PMA / Ionomycin (positive control) (PMA 2 ng/mL; ionomycin 1 μg/mL; Merck, Darmstadt, Germany) and 10 µg /ml LPS (Merck, Darmstadt, Germany ) at 37°C ,5% CO2 for 6-7 hours. After 1 hour of incubation, 1 μg/mL brefeldin A (BD Pharmingen, USA) will be added to all the wells. After incubation, cells will be surface stained for 25-30 minutes with anti-CD3FITC, anti-CD8BV421 and anti-CD4 PE/cyanine5.5 (Cy5) followed by 10 minutes permeabilization with 100 µL of permeabilising solution( BD Biosciences, USA) and will be washed twice with 500 µL 1x cytoperm. After washing, cells will be stained for intracellular expression of IL-2, IFN- γ and IL-17 with anti-IL2 APC, anti-IFN-γ PE, anti-IL-17 PE- Cy7 (BD Biosciences and Pharmingen, USA) and will be incubated for 25-30 minutes followed by washing with PBS and fixing the cells in 0.1 % PFA before acquiring on a BD Verse flow cytometer. Data will be analyzed using FlowJo software version 10.

Switching of monocyte Phenotype and functionality:

The blood samples at baseline (pre first dose), day 28 (4 weeks/28 days after first dose and just before second dose), 8 weeks (or 4 weeks after second dose), 16 weeks (or 12 weeks after second dose), 28 weeks (or 24 weeks after second dose), 40 weeks (or 36 weeks after second dose) and 52 weeks ( or 48 weeks after second dose) Vaccine will induce an increase in proinflammatory cytokine production, which is dependent on trained immunity in innate immune cells. We will characterize the phenotype and functionality of monocytes before vaccination and after vaccination using flowcytometric analysis.

Those who are fully immunized and still developing clinical Covid 19 infection will be grouped together and immunological profile will be studied.

ELIGIBILITY:
Inclusion Criteria:

The following patients will be enrolled in the study under Group 1:

* Age greater than and equal to 18 years
* Evidence of liver cirrhosis established during the clinical investigations and/or hospital stay, as evidenced by clinical, endoscopic, radiological and/or histological criteria.
* Baseline Negative SARS-COV19 IgG neutralizing antibodies

The following patients (healthy controls) will be enrolled in the study:

* Age greater than and equal to 18 years
* Baseline Negative SARS-COV19 IgG neutralizing antibodies
* No previous COVID-19 infection
* No major respiratory, cardiac comorbid illnesses or malignancy or immunosuppressed state

Exclusion Criteria:

* Planned receipt of any vaccine other than the study intervention within 30 days before and after each study vaccination with the exception of the licensed seasonal influenza vaccination and the licensed pneumococcal vaccine. Participants will be encouraged to receive this vaccination at least 7 days before or after their study vaccine.
* Prior or concomitant vaccine therapy for COVID-19
* ICU patients
* Hemodynamically unstable patients, shock
* Significant encephalopathy, acute kidney injury
* Documented or suspected sepsis including chest infection
* ACLF (Acute on Chronic Liver Failure)
* Significant cardiac or respiratory co-morbidities
* Known allergy to vaccination
* Prior receipt of an investigational or licensed vaccine likely to impact on interpretation of the trial data (e.g. Adenovirus vectored vaccines, any coronavirus vaccines).
* History of allergic disease or reactions likely to be exacerbated by any component of the AZD1222 (Covishield) vaccine.
* Any history of angioedema.
* Any history of anaphylaxis.
* Pregnancy, lactation or willingness/intention to become pregnant during the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Currently or in last 3 weeks have: fever/cough/sorethroat/rhinorrhea/hemoptysis/breathlessness/chest pain/myalgia/nausea/vomiting/diarrhea/abdominal pain/loss of taste

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-03-19 (Estimated); Study Completion 2022-03-19 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of AZD1222(Covishield) (2 doses) in patients with liver cirrhosis as measured by proportion of patients with presence of antibodies titres compared with the control group. | 6 months
To evaluate the safety/tolerability of AZD1222(Covishield) (2 doses) in patients with liver cirrhosis as measured by comparison of safety profile of AZD1222 (Covishield) in both the groups | 6 months
  Safety/tolerability will be assessed by collecting the adverse event data,events of decompensation and new onset of COVID 19 infection by RTPCR.

SECONDARY OUTCOMES:
To study the profile of immune cells after vaccination. | 1 year
  Immune cells profile SARS CoV2 serum IgG Levels, Primary IFN-γ ELISPOT assay,CD4,CD8 etc.
To study the profile of cytokine signatures after vaccination. | 1 year
  cytokine signatures are IL-2,IL-17,TNF alpha,IL-6
The proportion of participants who have a post-treatment response (negative at baseline to positive post treatment with study intervention) for SARS-CoV-2 Nucleocapsid antibodies over time. | 1 year
The incidence of the first case of SARS-CoV-2 RT-PCR-positive symptomatic illness for a participant occurring at or after 15 days post second dose of study intervention using criteria from the CDC. | 1 year
The incidence of SARS-CoV-RT-PCR-positive severe or critical symptomatic illness occurring 15 days or more post second dose of study intervention. | 1 year
Incidence of adverse events | 28 days
Incidence of serious adverse events, medically attended adverse events, and adverse events of special interest. | Day 1 post Treatment
Incidence of serious adverse events, medically attended adverse events, and adverse events of special interest. | Day 7 post Treatment
Incidence of serious adverse events, medically attended adverse events, and adverse events of special interest. | Day 30 post Treatment
Incidence of local and systemic solicited adverse events. | Day 7 post treatment
Determine the rate of new SARS-CoV2 infections, including the mutant strains. | 1 year
To determine the clinical severity of new SARS-CoV2 infections, including that of mutant strains. | 1 year
  Clinical severity is determined by new onset of Pneumonia, Respiratory failure, and need of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided